CLINICAL TRIAL: NCT06889194
Title: Knowledge, Attitude and Barriers of Egyptian and Sudanese Dentists in Providing Oral Health Care to Geriatric Patients: a Cross-sectional Study
Brief Title: Knowledge, Attitude and Barriers of Egyptian and Sudanese Dentists in Providing Oral Care to Geriatric Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Abdulbagi Abdulhalim Mohammed, Knowledge, Attitude and Barriers of Egyptian and Sudanese Dentists in Providing Oral Health Care to Geriatric Patients: A Cross-sectional Study, Cairo University
Other Study IDs: Esraa Abdulbagi 14422022412792
Record Dates: First submitted 2025-03-07; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Knowledge, Attitude and Barriers of Egyptian and Sudanese Dentists in Providing Oral Health Care to Geriatric Patients
Keywords: knowledge, attitudes, and barriers of Egyptian and Sudanese dentists - Geriatric patient-
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study (Cross sectional study) is to assess the level of knowledge of Egyptian and Sudanese dentists about the oral health care needs of geriatric patients and to evaluate the attitude towards treating geriatric patients and barriers in providing care.

The data collection by validated questionnaires. The Dentists would fill out structured surveys addressing their knowledge, attitudes, and perceived barriers regarding geriatric dental care.

ELIGIBILITY:
Inclusion Criteria:

* Post graduated Sudanese and Egyptian Dentists currently practicing in Egypt and Sudan
* Experience: Dentists who have been practicing for at least 1 year to ensure they have enough experience to have formed opinions and practices regarding geriatric care.
* Age: 20-60 years

Exclusion Criteria:

* • Dentists Not Providing Geriatric Care: Dentists who exclusively work with Paediatric and do not treat elderly populations will be excluded.

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Gender Based: Yes — Sudanese and Egyptian dentists
Study Population: Post graduated Sudanese and Egyptian Dentists currently practicing in Egypt and Sudan
  * Experience: Dentists who have been practicing for at least 1 year to ensure they have enough experience to have formed opinions and practices regarding geriatric care.
  * Age: 25-60 years
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge, Attitude and Barriers of Egyptian and Sudanese Dentists in Providing Oral Health Care to Geriatric Patients: A Cross-sectional Study | from April 2025 to December 2026
  primary outcome: knowledge about geriatric oral health. Measured through a validated questionnaire (Madunic et al., 2021). Includes categories on demographics, opinion, knowledge, attitudes, and barriers.
  Source of Data:
  Responses to a validated questionnaire administered to Egyptian and Sudanese dentists.
  Methods of Assessment (Measurement):
  * Self-reported questionnaire with Likert-scale responses.
  * Questions covering demographics, knowledge, attitudes, and barriers.
  Comparability of Assessment Methods:
  The same questionnaire was used for all participants, ensuring uniformity.

SECONDARY OUTCOMES:
Knowledge, Attitude and Barriers of Egyptian and Sudanese Dentists in Providing Oral Health Care to Geriatric Patients: A Cross-sectional Study | from April 2025 to December 2026
  secondary outcome: Attitude towards treating geriatric patients and barriers in providing care
  Methods of Assessment (Measurement):
  - Self-reported questionnaire with Likert-scale responses.

IPD SHARING:
Plan to Share IPD: No